CLINICAL TRIAL: NCT03650335
Title: Effect of Two Different Volumes of Bupivacaine 0.25% Used in Ultrasound-guided Erector Spinae Plane (ESP) Block on Dermatome Spread: A Volume Study
Brief Title: Effect of Bupivacaine in Ultrasound-guided Erector Spinae Plane
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Celaleddin Soyalp, Assist .Prof., Yuzuncu Yil University
Other Study IDs: ESP
Record Dates: First submitted 2018-08-25; First posted 2018-08-28 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: Thoracotomy
Keywords: erector spine plan block; postoperative opioid consumption; thoracotomy; analgesia; anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group I: with a total of 20 mL 0.25% bupivacaine injection to be administered
- group II: with a total of 30 mL 0.25% bupivacaine injection to be administered

SUMMARY:
To investigate the effect of two different volumes of bupivacaine 0.25% used in ultrasound-guided erector spinae plane (ESP) block on dermatome spread and postoperative analgesia in patients undergoing unilateral thoracotomy

DETAILED DESCRIPTION:
The study will have a double-blind design and will be conducted after obtaining an approval from the local ethics committee. The study will include 50 patients planned for thoracotomy, aged 18-65 years with an ASA score of I-II. The patients will be randomized by sealed tender and will be divided into 2 groups with 25 patients each. Patients that will be transferred to the intensive care unit (ICU) intubated after the surgery, patients with a body mass index of 35 or over, patients detected with infection in the intervention site, patients with hematological diseases, patients with a known allergy to local anesthetics, patients that will not provide a written or verbal consent, pregnant patients, and patients with an ASA score of III or IV will be excluded from the study. All the patients will undergo physical examination and their laboratory parameters will be evaluated one day prior to the procedure. Moreover, on the same day, each patient will be informed about dermatome testing (hot/cold), pain prick test (pain test), and pain pump set. Age, body height and weight, duration of block, and duration of surgery will be recorded for each patient

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective thoracotomy
* Aged 18-65 years
* ASA score of I and II

Exclusion Criteria:

* Patients that will be transferred to the intensive care unit (ICU) intubated after the surgery,
* Patients with a body mass index of 35 or over,
* Patients detected with infection in the intervention site,
* Patients with hematological diseases,
* Patients with a known allergy to local anesthetics,
* Patients that will not provide a written or verbal consent,
* Pregnant patients
* Patients with an ASA score of III or IV will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracotomy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | First 24 hours total opioid consumption
  Total opioid consumption as microgram/kg will be assessed in 24 hour surgery

CONTACTS AND LOCATIONS:
Overall Officials: celaleddin soyalp, Study Chair — Yuzuncu Yil University Dursun Odabas Medical School Anesthesiology and Reanimation Department Van, Turkey
Locations (1):
- Celaleddin Soyalp, Van, Turkey (Türkiye)